CLINICAL TRIAL: NCT04569955
Title: Knowledge and Perception of Clinical Trial Participation in Breast Cancer Female Patients in Egypt, a Cross Sectional Study
Brief Title: Knowledge and Perception of Clinical Trial Participation in Breast Cancer Patients in Egypt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hagar Elghazawy, Lecturer of clinical oncology, Ain Shams University
Other Study IDs: FMASU R61/2020
Record Dates: First submitted 2020-07-07; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer; Clinical Trials
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Knowledge and perception of clinical trial participation — This study aims to get a current picture of the patients' knowledge and perception of clinical trial participation in Breast cancer female patients in Egypt, as an example to Low/Middle income countries

SUMMARY:
* Clinical trials are essential to translate new therapy concepts or rather any intervention into the medical routine. Beside the well designed trial protocol, the success of clinical trials depends on patient recruitment and participation.
* This study aims to get a current picture of the patients' knowledge and perception of clinical trial participation in Breast cancer female patients in Egypt, as an example to Low/Middle income countries.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer patients

Exclusion Criteria:

* Patients who refuse participation

Max Age: 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: -Egyptian female Breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of breast cancer patients who accept to participate in clinical trials | 1 year

SECONDARY OUTCOMES:
The barriers for participation in clinical trials | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hagar Elghazawy, Principal Investigator — Ain shams university, faculty of medicine
Locations (1):
- Ain shams university, faculty of medicine, Cairo, Select, Egypt

IPD SHARING:
Plan to Share IPD: No